CLINICAL TRIAL: NCT05463861
Title: Lemborexant in Delayed Sleep Phase Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Emmanuel Mignot, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 59441
Record Dates: First submitted 2021-09-20; First posted 2022-07-19 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Delayed Sleep Phase Syndrome
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — lemborexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lemborexant (Active Comparator): Patients receive Lemborexant 5mg for 7 days and may be dose adjusted to 10mg. Patients continue to take Lemborexant 5mg or 10 mg for an additional 7 days.
  Interventions: Drug: Lemborexant
- Placebo (Placebo Comparator): Patients receive placebo to match Lemborexant for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lemborexant — Lemborexant tablet administered orally once daily.
  Other Names: dayvigo®
  Arms: Lemborexant
Drug: Placebo — Placebo to match Lemborexant tablet administered orally once daily.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate whether Lemborexant is more effective than placebo in shortening sleep onset latency in patients with delayed sleep phase syndrome (both type 1 and type 2). This will be tracked using sleep logs as well as actigraphy.

In this 2-year study, we will examine if Lemborexant administered 5-10 mg nightly taken at desired bedtime (at least 2 hours prior to self-reported sleep onset habitual time) can improve the symptoms of Delayed Sleep Phase Syndrome.

DETAILED DESCRIPTION:
Delayed sleep phase syndrome (DSPS) is a disorder in which a person's sleep is delayed by two hours or more beyond what is considered an acceptable or conventional bedtime. The delayed sleep then causes difficulty in being able to wake up at the desired time.

In DSPS, bedtime is shifted later than the general population such that individuals have difficulty getting enough sleep to meet their sleep needs before they have to get up for their daytime obligations (work, school, childcare, etc.). As a result, patients experience daytime impairment, including daytime sleepiness and cognitive impairment. DSPS, if maintained in adulthood, is associated with numerous deleterious health effects, although causality is not well established. Two phenotypes of DSPS are recognized depending on the phase of entrainment: one with a late phase and normal phase angle (non-circadian) and other with a late phase and abnormal phase angle (circadian). The differentiation of these two phenotypes is theoretical: a mixed situation may be involved in some cases and the exact pathophysiology of each subtype is still controversial.

In theory, however, separating the sample into these two subtypes is likely important to predict short- and long-term responses to orexin antagonists in DSPS.

Lemborexant is one of the dual orexin receptor antagonists on the US market. The purpose of this study is to examine if lemborexant administered 5 to 10 mg nightly, taken at desired bedtime (at least 2 hours prior to self-reported sleep onset time), can improve the symptoms of Delayed Sleep Phase Syndrome both in the circadian and non-circadian phenotypes. The phenotypes will be recruited in 1:1 proportion.The effect of lemborexant will be analyzed based on the collection of information from actigraphy watches, sleep diaries, and sleep scales. The total participation time involved in this study will be approximately 6 weeks (2 weeks of baseline assessment followed by 2-weeks of treatment/placebo, and 2 weeks post-treatment).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Diagnosed with delayed sleep phase syndrome (DSPS) meaning that:

   1. Sleep is delayed by two hours or more beyond what is considered an acceptable or conventional bedtime for the subject (their desired bedtime).
   2. Subjects not able to fall asleep if trying to sleep before the later bedtime;
   3. This is interfering with their wishes/having social impact.
3. Concomitant medications will be allowed, though dosages will be required to remain fixed throughout participation in the study.
4. The participant also needs to be willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Clinically significant depression (PHQ-9 score of 10 or more), anxiety disorder (GAD-7 score of 10 or more), substance use disorder, any other sleep disorder (assessed by the Alliance Sleep Questionnaire- ASQ), or any medical disorder/therapy that could interfere with the trial (this will be verified through interview and analysis of the ASQ).
2. Use of medications with significant effects on sleep-wake function (insomnia therapies, stimulants)- unless they are discontinued at least 5 half-lives prior to study participation. Non-sedative antidepressants or SSRI will be allowed if at a stable dose in the absence of concomitant severe depression or severe anxiety.
3. Use of CYP3A inhibitors and CYP3A inducers, at least 1 week (or five half-lives, whichever is longer) prior to the first day of the baseline phase.
4. Pregnancy (verified by urine pregnancy test on visits 1, 2, and 3) or plan to become pregnant in the next 3 months or currently breastfeeding.
5. Shift workers or subjects working unusual hours.
6. Any risk of suicide within 6 months of screening period or throughout the trial (accessed by the Investigator and by the C-SSRS questionnaire).
7. Transmeridian travel across more than 3 time zones 4 weeks prior to the screening phase.
8. Transmeridian travel across more than 2 time zones during this trial (including the screening phase).
9. Having a positive drug test or being unwilling to refrain from using illegal drugs or marijuana during this trial.
10. Any clinically abnormal symptom or organ impairment found by medical history at Screening or Baseline and physical examinations, vital signs, ECG findings, or laboratory test results that require medical treatment.
11. Impaired liver function (values for enzymes aspartate transaminase (AST) and alanine transaminase (ALT) > 1.5 times the Upper Limit of Normal).
12. Known to be human immunodeficiency virus positive.
13. Has a QT interval corrected using Fridericia's formula interval (QTcF interval) >450 ms demonstrated on repeated ECGs (repeated only if initial ECG showed corrected QT interval (QTc) >450 ms) at Screening or Baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in actigraphy sleep latency onset | From 2 weeks prior to randomization to 4 weeks post randomization
  Sleep latency is the time from laying down until falling asleep. Actigraphy data obtained using Axivity- AX6.

SECONDARY OUTCOMES:
Change in Epworth Sleepiness Scale (ESS) | From randomization to 4 weeks post randomization
  This is a scale to evaluate daytime sleepiness. Range from 0 to 24 points (higher scores mean more sleepiness).
Change in Karolinska Sleepiness Scale (KSS) | From randomization to 4 weeks post randomization
  Self-report for daytime sleepiness with 1 being extremely alert and 10 being extremely sleepy, can't keep awake.
Change in sleep diary derived sleep onset latency | From 2 weeks prior to randomization to 4 weeks post randomization
  Sleep latency is the time from laying down until falling asleep as estimated by patient in dairy.
Sleep Regularity Index | From 2 weeks prior to randomization to 4 weeks post randomization
  Sleep Regularity Index is defined as the percentage probability of a person being asleep (or awake) at any two time points 24 hours apart. Actigraphy data obtained using Axivity- AX6.
Change in actigraphy derived total sleep time | From 2 weeks prior to randomization to 4 weeks post randomization
  Actigraphy data obtained using Axivity- AX6.
Change in sleep diary derived total sleep time. | From 2 weeks prior to randomization to 4 weeks post randomization
  Estimated by patient in dairy.
Change in mean actigraphy derived wake time | From 2 weeks prior to randomization to 4 weeks post randomization
  Wake time is total time awake over night after sleep onset. Actigraphy data obtained using Axivity- AX6.
Change in mean sleep diary derived wake time | From 2 weeks prior to randomization to 4 weeks post randomization
  Wake time is total time awake over night after sleep onset as estimated by patient in dairy.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mignot, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Univeristy, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No